CLINICAL TRIAL: NCT05157009
Title: Immediate Implants in Damaged Sockets With Simultaneous Bone Reconstruction vs. Immediate Implants in Intact Sockets and no Reconstruction
Brief Title: Immediate Implant Outcomes With and Without Bone Augmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Verdugo, Fernando, DDS (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VerdugoF
Record Dates: First submitted 2021-11-08; First posted 2021-12-14 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Tooth Loss; Bone Loss, Alveolar; Dental Diseases; Dental Trauma
Keywords: immediate dental implant; dental implant; bone regeneration; peri-implantitis
MeSH Terms: conditions — Tooth Loss; Alveolar Bone Loss; Stomatognathic Diseases; Peri-Implantitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate implant placement without reconstruction (Other): Immediate implant placement after tooth extraction
  Interventions: Procedure: implant placement
- Immediate implant placement with reconstruction (Other): Immediate implant placement and simultaneous bone reconstruction after tooth extraction
  Interventions: Procedure: implant placement

INTERVENTIONS:
Procedure: implant placement — autogenous bone reconstruction of damaged socket & simultaneous implant placement
  Other Names: bone reconstruction

SUMMARY:
To evaluate immediate implant placement feasibility and esthetic outcomes in severely damaged sockets that received simultaneously bone reconstruction (cortical bone shield) and implant placement versus intact sockets that needed no reconstruction and had immediate implant placement.

DETAILED DESCRIPTION:
The present clinical trial aims at demonstrating facial bone regeneration on sites that presented large buccal bone dehiscences & vertical bone loss and evaluate the feasibility of performing simultaneous bone augmentation and implant placement, comparing the outcomes with sites that had intact sockets that did not require reconstruction. A secondary objective was to evaluate pink esthetics and marginal bone levels at final follow-up.

ELIGIBILITY:
Inclusion Criteria:

* individuals 20 Years and older
* Patients requiring single implants to replace missing teeth to restore masticatory function and esthetics.
* ASA1 or ASA2 (American Society of Anesthesiologists)
* Healthy individuals with good oral hygiene and motivation
* No systemic uncontrolled diseases
* Not taking drugs known to modify bone metabolism

Exclusion Criteria:

* Individuals with untreated & generalized severe periodontitis
* Smokers (>5 cigarettes/day)
* Poor oral hygiene
* Diabetes (HbA1C >6.5% as cutoff value)
* Uncontrolled cardiovascular disease
* Poor overall health (ASA IV)

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate implant placement feasibility & success rate at 12 months | 12 months
  evaluate implant success following Karoussis et al. success criteria
Number of individuals with low pink esthetic outcomes as assessed by pink esthetic scores (PES) | 12 months
  pink esthetics scores (PES) as proposed by Belser et al. Values 0-10 were 10 is the best esthetic outcome.

SECONDARY OUTCOMES:
Implant transparency: clinical presence or absence | 12 months
  Visual evaluation of facial mucosal implant transparency at 12 months: positive or negative
Number of participants with >0.2mm of marginal bone levels | 12 months
  evaluate radiographic marginal bone levels at 12 months with >0.2mm of bone loss
Band of keratinized tissue: clinical presence or absence | 12 months
  evaluate the presence of facial keratinized tissue on the implant sites >2 or <2mm

CONTACTS AND LOCATIONS:
Overall Officials: Verdugo, PhD, Principal Investigator — Verdugo, Fernando, DDS
Locations (1):
- FV, DDS,Corp, San Gabriel, California, United States